CLINICAL TRIAL: NCT05466149
Title: A Phase 2, Multicenter, Open-Label Study to Assess the Efficacy and Safety of Furmonertinib in Patients With Locally Advanced or Metastatic Non-Small Cell Lung Cancer (NSCLC) With Epidermal Growth Factor Receptor (EGFR) Exon 20 Insertion Mutations
Brief Title: Efficacy and Safety of Furmonertinib in Patients With Locally Advanced or Metastatic NSCLC With EGFR Exon 20 Insertion
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Allist Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FURMO-003
Record Dates: First submitted 2022-07-14; First posted 2022-07-20 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-03

CONDITIONS: NSCLC
MeSH Terms: interventions — aflutinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Furmonertinib 240mg QD (Experimental): Treating patients of locally advanced or metastatic NSCLC with EGFR exon 20 insertions who have progressed during or after platinum-based chemotherapy.
  Interventions: Drug: Furmonertinib

INTERVENTIONS:
Drug: Furmonertinib — 240mg QD on a continuous dosing schedule.
  Other Names: AST2818

SUMMARY:
This is a Phase 2, Multicenter, Open-Label Study to Assess the Efficacy and Safety of Furmonertinib in Patients with Locally Advanced or Metastatic Non-Small Cell Lung Cancer (NSCLC) with Epidermal Growth Factor Receptor (EGFR) Exon 20 Insertion Mutations.

The study plans to enroll approximately 100 patients from approximately 70 sites. Patients are locally advanced or metastatic NSCLC with EGFR exon 20 insertions who have progressed during or after platinum-based chemotherapy. Furmonertinib Mesilate will be treated 240 mg QD until disease progression or unacceptable toxicity.

Primary endpoint is ORR. Secondary endpoints include DOR, DCR, DepOR, PFS, OS, CNS ORR, CNS DOR, CNS PFS, safety and the PK profile of Furmonertinib Mesilate and its metabolites (AST5902).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at time of signing Informed Consent Form
* Histologically or cytologically documented, locally advanced or metastatic NSCLC not amenable to curative surgery or radiotherapy
* Documented validated results from local or central testing (as designated by the Sponsor) of blood or tumor tissue confirming the presence of an EGFR exon 20 insertion mutation
* Documented radiologic progression on or after prior platinum-based chemotherapy (with or without anti-PD1/PD-L1 agents) in the locally advanced or metastatic setting
* Documented radiologic disease progression during or after the last systemic anticancer therapy before the first dose of furmonertinib
* Measurable disease per RECIST v1.1
* ECOG performance status of 0 or 1
* Life expectancy of ≥ 12 weeks
* Patients with CNS metastases are eligible, provided they meet all of the following criteria: Measurable disease outside the CNS; No ongoing requirement for corticosteroids as therapy for CNS metastases, with corticosteroids discontinued for ≥ 2 weeks prior to enrollment; No ongoing symptoms attributed to CNS metastases; No active CNS metastases or spinal cord compression (i.e., progressing or requiring anticonvulsants or corticosteroids for symptomatic control); No evidence of interim CNS disease progression between the completion of CNS-directed therapy and the screening radiographic study; Time since whole brain radiation therapy (WBRT) is ≥ 21 days prior to first dose of study treatment, time since stereotactic radiosurgery (SRS) is ≥ 7 days prior to first dose of study treatment, or time since surgical resection is ≥ 28 days
* Adequate hematologic and organ function within 14 days prior to initiation of study treatment
* For women of childbearing potential or men who are not surgically sterile: Agreement to remain abstinent or use contraception, and agreement to refrain from donating eggs or sperm

Exclusion Criteria:

* Prior treatment with any EGFR-targeting agents (e.g., EGFR tyrosine kinase inhibitors [TKIs], monoclonal antibodies, or bispecific antibodies).
* More than 3 prior systemic anticancer therapy regimens for locally advanced or metastatic NSCLC
* Inability or unwillingness to swallow pills
* Severe acute or chronic infections
* Previous interstitial lung disease (ILD), drug-induced ILD, radiation pneumonitis requiring steroid therapy; or having the clinical manifestations of suspected ILD
* History of or active clinically significant cardiovascular dysfunction
* Mean resting corrected QT interval (QTc) > 470 msec, obtained from triplicate ECGs, using the screening clinic ECG machine derived Fridericia's formula (QTcF) value
* Clinically significant prolonged QT interval or other arrhythmia or clinical status considered by investigators that may increase the risk of prolonged QT interval (e.g., complete left bundle branch block, degree III atrioventricular block, second-degree heart block, PR interval > 250 msec, congenital long QT syndrome, family history of long QT syndrome, or unexplained sudden death under 40 years of age in first-degree relatives, serious hypokalemia, heart failure) or current use of the drugs that may lead to prolonged QT interval.
* AEs from prior anticancer therapy that have not resolved to Grade ≤ 1 except for alopecia, vitiligo, endocrinopathy managed with replacement therapy, or Grade ≤ 2 peripheral neuropathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-09-27 (Actual); Primary Completion 2025-06-27 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
ORR, Objective Response Rate | Approximately 7.5 months following the last patient enrolled
  Percentage of patients with a confirmed CR or PR relative to the total number of patients.

SECONDARY OUTCOMES:
DOR, Duration of response | Approximately 7.5 months following the last patient enrolled
  Time from first documented evidence of confirmed CR or PR until the first documented evidence of disease progression or death, whichever occurs earlier
DCR, Disease control rate | Approximately 7.5 months following the last patient enrolled
  Proportion of patients with CR, PR, or SD
Depth of response | Approximately 7.5 months following the last patient enrolled
  Maximum reduction in BICR and investigator assessment using RECIST v1.1 compared to baseline
PFS, Progression Free Survival | Approximately 7.5 months following the last patient enrolled
  Time from first dose date to the first occurrence of disease progression, or death from any cause, whichever occurs first
OS, Overall Survival | Approximately 3 years following the last patient enrolled
  Time from first dose to death from any cause
CNS ORR, CNS DOR, CNS PFS | Approximately 7.5 months following the last patient enrolled
  Evaluated by BICR per modified RECIST criteria in patients with CNS lesion(s) on baseline brain scan
Adverse Events | Until 28 days from the last dose of study drugs or initiation of a new anticancer treatment
  Incidence and severity of adverse events, with severity determined according to National Cancer Institute Common Terminology Criteria for Adverse Events, Version 5.0 (NCI CTCAE v5.0).
Maximum Plasma Concentration [Cmax] | Approximately 7.5 months following the last patient enrolled
  Plasma concentrations of furmonertinib and its major metabolite (AST5902) at specified time points
Minimum Plasma Concentration [Cmin] | Approximately 7.5 months following the last patient enrolled
  Plasma concentrations of furmonertinib and its major metabolite (AST5902) at specified time points

CONTACTS AND LOCATIONS:
Locations (1):
- Jilin Province Cancer Hospital, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No